CLINICAL TRIAL: NCT07183384
Title: The Effectiveness of Mesenchymal Stem Cell-Derived Exosome Therapy in Improving Endothelial Dysfunction in Postpartum Mothers With a History of Preeclampsia
Brief Title: MSC Exosome Therapy for Post-Preeclampsia Endothelial Dysfunction
Acronym: EXITPE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Dr. Hasan Sadikin General Hospital, Bandung, Indonesia (Unknown); Dr Cipto Mangunkusumo General Hospital (Other); Dr. Sardjito Hospital, Yogyakarta (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OBGY-202508.01
Record Dates: First submitted 2025-09-02; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Preeclampsia; Postpartum; Endothelial Injury; Exosome Multiomics; Cell Therapy
Keywords: Preeclampsia; Postpartum; Stem Cell; Exosome; Cell Therapy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled clinical trial with parallel group design. Participants will be randomized 1:1 to receive either MSC-derived exosomes or placebo (sterile saline solution). Both groups will be followed for the same duration with identical assessment schedules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC-derived Exosome Therapy (Experimental): Participants receive Intravenous or Intramuscular MSC-derived exosomes.
  Interventions: Biological: Mesenchymal Stem Cell-Derived Exosomes
- Saline/Placebo (Placebo Comparator): Participants receive Intravenous or Intramuscular sterile saline solution
  Interventions: Other: Placebo (Sterile Saline Solution)

INTERVENTIONS:
Biological: Mesenchymal Stem Cell-Derived Exosomes — Mesenchymal stem cell-derived exosomes isolated from adipose-derived stem cells (ASC). The exosomes contain bioactive molecules including microRNAs (particularly miR-126-3p), proteins, and lipids that promote endothelial repair and regeneration. The product is manufactured under GMP conditions and administered as a single Intravenous or Intramuscular infusion.
  Other Names: MSC-Exos; Fetal stem cell exosomes
  Arms: MSC-derived Exosome Therapy
Other: Placebo (Sterile Saline Solution) — Sterile saline solution (0.9% sodium chloride) administered Intravenous or Intramuscular as placebo control. The volume and administration method are identical to the active treatment to maintain blinding.
  Other Names: Normal saline; 0.9% sodium chloride
  Arms: Saline/Placebo

SUMMARY:
---

Why Is This Study Being Done?

Women who have preeclampsia during pregnancy face a much higher risk of heart disease later in life. Preeclampsia is a serious pregnancy condition that causes high blood pressure and damages blood vessels. Even after the baby is born, the blood vessels do not fully heal on their own, which can lead to heart problems/cardiovascular years later.

This study tests whether a new treatment called exosomes can help repair damaged blood vessels in women who had preeclampsia. Exosomes are tiny particles that come from stem cells and contain healing substances that may help blood vessels work better.

---

What Will Happen in This Study?

This study will include 80 women who recently gave birth and had preeclampsia during their pregnancy. Half of the women will receive the exosome treatment through an IV, and half will receive a placebo (a substance with no active treatment).

---

What Will Participants Need to Do?

Participants will:

* Have blood tests and other health checks
* Receive one treatment through an IV
* Return for follow-up visits at 1 week after treatment
* Have tests to check how well their blood vessels are working

Who Can Join This Study?

Women who:

* Recently gave birth (within 1-2 weeks)
* Had preeclampsia during their last pregnancy
* Are healthy enough to participate
* Can give permission to join the study

What Are the Possible Benefits and Risks?

The treatment may help repair blood vessel damage and reduce the risk of future heart disease. The exosome treatment appears to be safe based on other studies, but like any medical treatment, there may be side effects.

---

How Long Will the Study Last?

The main treatment happens during one visit, with follow-up visits for 1 week to check on participants' health and see if the treatment is working.

This research may lead to new ways to protect women's heart health after pregnancy complications.

DETAILED DESCRIPTION:
---

Background and Rationale

Preeclampsia affects 3-5% of pregnancies globally and represents a severe pregnancy-specific syndrome characterized by widespread maternal endothelial dysfunction. The pathophysiology involves abnormal trophoblast invasion leading to placental ischemia. Beyond immediate perinatal risks, preeclampsia carries devastating long-term cardiovascular consequences, with women experiencing a four-fold increased risk of heart failure, a 2.5-fold increased risk of coronary heart disease, and a two-fold increased risk of stroke and cardiovascular death. Moreover, post-cesarean postpartum mothers with a history of preeclampsia face particularly elevated risks, with cesarean delivery increasing postpartum preeclampsia risk by two- to seven-fold compared to vaginal delivery. This increased risk stems from altered hemodynamics, surgical stress responses, and compromised vascular integrity following cesarean procedures.

---

Scientific Innovation

This study represents a paradigm shift from symptomatic management to active regenerative therapy using mesenchymal stem cell-derived exosomes (MSC-Exos). MSC-Exos offer several advantages over traditional approaches: natural tropism for vascular tissues, multi-pathway targeting capabilities, reduced immunogenicity compared to cell-based therapies, and superior circulation stability. Recent systematic reviews demonstrate favorable safety profiles with a low incidence of serious adverse events (0.7%).

---

Intervention Details

Participants will receive a single intravenous or intramuscular dose of MSC-derived exosomes obtained from fetal adipose stem cells (ASC), produced under Good Manufacturing Practice (GMP) conditions. The exosomes contain bioactive cargo including growth factors, cytokines, proteins, and therapeutic microRNAs (particularly miR-126-3p) that mediate intercellular communication and tissue repair. Control participants will receive sterile saline solution of identical volume via the same route.

---

Biomarker Strategy

The study employs miR-126-3p as the primary biomarker based on its exceptional diagnostic performance for endothelial dysfunction. miR-126-3p demonstrates high sensitivity (85.71%) and specificity (81.82%) with an area under the curve (AUC) of 0.792 for detecting endothelial dysfunction. This microRNA serves dual roles as both a pathological mediator and therapeutic target, making it ideal for monitoring treatment response. miR-126-3p is significantly downregulated in preeclampsia and directly regulates key angiogenic pathways including PI3K/AKT and MAPK/ERK signaling.

---

Mechanistic Rationale

MSC-derived exosomes promote endothelial repair through multiple complementary mechanisms:

* Anti-inflammatory effects by promoting M2 macrophage polarization and reducing pro-inflammatory cytokines (IL-1β, IL-6, TNF-α).
* Angiogenic promotion through delivery of pro-angiogenic factors including VEGF, VEGFR-2, and specific microRNAs.
* Anti-apoptotic activity protecting endothelial cells via regulation of Bcl-2/Bax/Caspase-3 pathways.
* Vascular barrier protection by maintaining intercellular junctions and preventing vascular permeability.

Clinical Assessment Protocol

The study incorporates comprehensive clinical monitoring including Hematology examination (Hemoglobin, MCV & MCHC, Hematocrit, Leukocyte, Platelets), Vital Signs Assessment (Blood Pressure, Respiratory Rate, Heart Rate), Edema assessment (Upper Extremity Edema, Lower Extremity Edema, Facial Edema), proteinuria evaluation, and Imaging Outcome (Pulsatility Index (PI), and Resistance Index (RI) Uterine Artery, Uterine Involusion)

---

Therapeutic Window and Follow-Up

The intervention targets the critical postpartum period (first-second week) when endothelial regeneration naturally occurs but may be compromised in preeclampsia patients. The 24-month follow-up period aligns with evidence suggesting therapeutic interventions during early postpartum may help reset long-term cardiovascular risk trajectories. This extended monitoring allows assessment of sustained therapeutic effects and long-term cardiovascular protection.

---

Statistical Considerations

Sample size calculation (n=40 per group) is based on power analysis with α=0.05 and 80% power, accounting for a 10% dropout rate. The study design incorporates interim analysis at 50% recruitment with predetermined safety stopping rules monitored by an independent Data Safety Monitoring Board.

---

Expected Clinical Impact

This study could establish a new therapeutic paradigm for postpartum care, shifting from reactive symptomatic management to proactive regenerative intervention. Success would provide the foundation for developing standardized exosome therapy protocols, potentially reducing long-term cardiovascular disease burden in high-risk postpartum populations, and contributing to improved maternal health outcomes with significant economic implications for healthcare systems.

---

Regulatory and Safety Framework

The study operates under comprehensive ethical oversight with approval from the institutional Health Research Ethics Committee. Safety monitoring includes comprehensive adverse event reporting protocols and predefined safety stopping criteria to ensure participant protection throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum
* Confirmed diagnosis of preeclampsia in the last pregnancy
* Postpartum period of first week and second week
* Able to provide informed consent

Exclusion Criteria:

* History of chronic hypertension prior to pregnancy
* Major cardiovascular disease history
* Active systemic infection
* Endothelial Injury history
* Active smoking status including vape, alcohol, drug addiction.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only biologically female participants who are postpartum mothers with a history of preeclampsia are eligible to participate in this study.
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Endothelial Function Biomarker (miR-126-3p) | Baseline and 1 week post-intervention
  Measure: Change in miR-126-3p expression levels from baseline to 1 week post-intervention.
  Method: RT-PCR analysis of blood samples. Unit: Fold change (relative expression). Scale Description: Continuous variable measured as fold change relative to baseline. Higher values indicate improved endothelial function. Normal range: 0.8-1.2 fold change. Values <0.8 indicate dysfunction.

SECONDARY OUTCOMES:
Systolic Blood Pressure | Baseline, first week, and 1 week post-intervention
  Measure: Change in systolic blood pressure from baseline. Unit: mmHg. Normal Range: 90-140 mmHg (postpartum). Values ≥140 mmHg indicate hypertension.
Diastolic Blood Pressure | Baseline, first week, and 1 week post-intervention
  Measure: Change in diastolic blood pressure from baseline.
  Unit: mmHg.
  Normal Range: 60-90 mmHg (postpartum). Values ≥90 mmHg indicate hypertension.
Hemoglobin Level | Baseline and 1 week post-intervention
  Measure: Change in hemoglobin concentration from baseline.
  Unit: g/dL.
  Normal Range: 11.0-15.0 g/dL (postpartum). Values <11.0 g/dL indicate anemia.
Hematocrit Level | Baseline and 1 week post-intervention
  Measure: Change in hematocrit percentage from baseline.
  Unit: Percentage (%).
  Normal Range: 33-45% (postpartum). Values <33% indicate anemia.
Leukocyte Count | Baseline and 1 week post-intervention
  Measure: Change in white blood cell count from baseline.
  Unit: cells/μL.
  Normal Range: 9,000-25,000 cells/μL (postpartum, elevated due to normal physiologic stress). Values >25,000 may indicate infection.
Platelet Count | Baseline and 1 week post-intervention
  Measure: Change in platelet count from baseline.
  Unit: cells/μL.
  Normal Range: 150,000-400,000 cells/μL. Values <150,000 indicate thrombocytopenia.
Mean Corpuscular Volume (MCV) | Baseline and 1 week post-intervention
  Measure: Change in mean corpuscular volume from baseline.
  Unit: femtoliters (fL).
  Normal Range: 80-100 fL. Values <80 fL indicate microcytic anemia; >100 fL indicate macrocytic anemia.
Mean Corpuscular Hemoglobin Concentration (MCHC) | Baseline and 1 week post-intervention
  Measure: Change in mean corpuscular hemoglobin concentration from baseline.
  Unit: g/dL.
  Normal Range: 32-36 g/dL. Values <32 g/dL indicate hypochromic anemia.
Proteinuria Level | Baseline and 1 week post-intervention
  Measure: Change in urine protein level from baseline using dipstick urinalysis.
  Unit: Dipstick protein scale (qualitative).
  Scale Description: Urine Dipstick Protein Scale:
  Negative/Trace: Normal (no significant proteinuria)
  1. (30 mg/dL): Mild proteinuria
  2. (100 mg/dL): Moderate proteinuria
  3. (300 mg/dL): Severe proteinuria
  4. (>2000 mg/dL): Very severe proteinuria
  Normal Range: Negative to Trace in postpartum period.
  Interpretation: Higher grades indicate worse proteinuria. Grades 2+ and above indicate clinically significant proteinuria requiring monitoring.
Uterine Artery Pulsatility Index (PI) | Baseline and 1 week post-intervention
  Measure: Change in Pulsatility Index of uterine artery measured by Doppler ultrasound.
  Unit: Ratio (dimensionless).
  Scale Description: Calculated as (peak systolic velocity - end diastolic velocity)/mean velocity. Normal postpartum range: 0.5-1.2. Higher values indicate increased vascular resistance.
Uterine Artery Resistance Index (RI) | Baseline and 1 week post-intervention
  Measure: Change in Resistance Index of uterine artery measured by Doppler ultrasound.
  Unit: Ratio (dimensionless).
  Scale Description: Calculated as (peak systolic velocity - end diastolic velocity)/peak systolic velocity. Normal postpartum range: 0.4-0.8. Higher values indicate increased vascular resistance.
Heart Rate | Baseline, first week, and 1 week post-intervention
  Measure: Change in heart rate from baseline.
  Unit: beats per minute (bpm).
  Normal Range: 60-100 bpm (postpartum may be slightly elevated 70-110 bpm). Values >110 bpm may indicate tachycardia.
Respiratory Rate | Baseline, first week, and 1 week post-intervention
  Measure: Change in respiratory rate from baseline
  Unit: breaths per minute
  Normal Range: 12-20 breaths per minute. Values >20 may indicate tachypnea.
Upper Extremity Edema Grade | Baseline and 1 week post-intervention
  Measure: Change in upper extremity edema grading from baseline.
  Unit: Grade on standardized scale.
  Scale Description: Postpartum Edema Grading Scale (0-4):
  Grade 0: No edema
  Grade 1: Mild pitting edema, barely perceptible
  Grade 2: Moderate pitting edema, clearly visible
  Grade 3: Severe pitting edema with obvious swelling
  Grade 4: Very severe pitting edema with marked deformity.
  Interpretation: Higher grades indicate worse edema. Grade 0-1 considered normal postpartum; Grades 2-4 indicate pathological edema.
Lower Extremity Edema Grade | Baseline and 1 week post-intervention
  Measure: Change in lower extremity edema grading from baseline.
  Unit: Grade on standardized scale.
  Scale Description: Postpartum Edema Grading Scale (0-4) - same as above.
  Interpretation: Higher grades indicate worse edema. Grade 0-1 considered normal postpartum; Grades 2-4 indicate pathological edema.
Facial Edema Grade | Baseline and 1 week post-intervention
  Measure: Change in facial edema grading from baseline.
  Unit: Grade on standardized scale.
  Scale Description: Postpartum Edema Grading Scale (0-4) - same as above.
  Interpretation: Higher grades indicate worse edema. Grade 0 considered normal postpartum; Grades 1-4 indicate pathological edema.
Uterine Involution Status | Baseline and 1 week post-intervention
  Measure: Assessment of uterine involution progress measured by uterine height.
  Unit: centimeters (cm) above symphysis pubis.
  Normal Range:
  Day 1 postpartum: At umbilicus (~12 cm)
  Day 7 postpartum: 7-9 cm above symphysis pubis
  Day 14 postpartum: 4-6 cm above symphysis pubis.
  Interpretation: Expected decrease of ~1 cm per day. Slower decrease may indicate subinvolution.

OTHER OUTCOMES:
Number of participants with clinically significant abnormal laboratory test results | Baseline to 7 days after last dose of exosomes.
  Number and percentage of participants with ≥1 clinically significant abnormal laboratory result after baseline. "Clinically significant" = laboratory value outside normal reference range and meeting pre-specified criteria in protocol (investigator-assessed clinically important change). Each participant counted once regardless of number of abnormal tests.

CONTACTS AND LOCATIONS:
Overall Officials: Akhmad Y Pramatirta, M.D., Ph.D, Principal Investigator — Dr. Hasan Sadikin Central General Hospital
Locations (1):
- Dr. Hasan Sadikin Central General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications from this study will be shared after de-identification, including biomarker data (miR-126-3p), clinical outcomes, safety parameters, and demographic data collected according to the study protocol. Sensitive information that could potentially re-identify participants will be excluded from shared datasets.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data and supporting documents will be available beginning 9 months and ending 60 months following article publication. This timeframe allows for completion of primary analyses and preparation of data for sharing while ensuring long-term availability for secondary research and meta-analyses.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for secondary research purposes including individual participant data meta-analyses. Requestors must have approval from an Institutional Review Board (IRB) or Independent Ethics Committee (IEC) and execute a data sharing agreement with Dr. Hasan Sadikin Central General Hospital. Proposals should be directed to akhmad.yogi@unpad.ac.id. Access will be granted for analyses that align with the study's scientific objectives and ethical considerations

REFERENCES:
- [Background] Vioretti, R., Khairani, A. F., Fauziah, P. N., & Hilmanto, D. (2018). An evaluation of soyghurt potential on tumor necrosis factor-α and soluble endoglin levels in preclampsia maternal serum-induced placental trophoblast cell in vitro. International Food Research Journal, 25(4), 1397-1402.
- [Background] Gurnadi, J. I., Mose, J. C., Handono, B., Fauziah, P. N., & Pramatirta, A. Y. (2015). Correlation between fms-Like tyrosine kinase-1 (sFlt-1) cell-free messenger RNA expression and fms-Like tyrosine kinase-1 (sFlt-1) protein level in severe preeclampsia and normal pregnancy. International Journal of Integrated Health Sciences, 3(2), 66-71.
- [Background] Pramatirta AY, Mose J, Effendi JS, Krisnadi SR, Anwar AD, Fauziah PN, Gurnadi JI, Rihibiha DD. Correlation between cell-free mRNA expressions and PLGF protein level in severe preeclampsia. BMC Res Notes. 2015 Jun 2;8:208. doi: 10.1186/s13104-015-1186-9. PMID 26032325